CLINICAL TRIAL: NCT00047775
Title: African-American Heart Failure Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nitromed (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: A-HeFT
Record Dates: First submitted 2002-10-18; First posted 2002-10-21 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-10

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — isosorbide-hydralazine combination

INTERVENTIONS:
Drug: BiDil

SUMMARY:
A placebo-controlled trial of BiDil added to standard therapy in African-American patients with heart failure.

DETAILED DESCRIPTION:
The overall objective is confirmation of BiDil's Safety and Efficacy in African-American (AFA) Patients with Moderate to Severe Symptomatic Heart Failure.

ELIGIBILITY:
* African American male or female 18 years or older.
* NYHA Class 3 & 4.
* Have either a resting LVEF less than or equal to 35% (by any method) or a resting LVIDD greater than 2.9 cm/m2 BSA (or greater than 6.5 cm) with LVEF less than 45% (by echocardiogram).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100
Dates: Start 2001-05; Study Completion 2004-08

CONTACTS AND LOCATIONS:
Overall Officials: Anne L. Taylor, M.D., Study Chair — University of Minnesota
Locations (7):
- United States (7):
  - Cooper Green Hospital, Birmingham, Alabama
  - Cardiology and Medicine Clinic, Little Rock, Arkansas
  - Howard University Hospital, Washington D.C., District of Columbia
  - Miami International Cardiology Consultants, Aventura, Florida
  - Boston Medical Center, Boston, Massachusetts
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Saint Vincents Hospital and Medical Center, New York, New York

REFERENCES:
- [Derived] Anand IS, Win S, Rector TS, Cohn JN, Taylor AL. Effect of fixed-dose combination of isosorbide dinitrate and hydralazine on all hospitalizations and on 30-day readmission rates in patients with heart failure: results from the African-American Heart Failure Trial. Circ Heart Fail. 2014 Sep;7(5):759-65. doi: 10.1161/CIRCHEARTFAILURE.114.001360. Epub 2014 Jun 26. PMID 24970468
- [Derived] Mitchell JE, Tam SW, Trivedi K, Taylor AL, O'Neal W, Cohn JN, Worcel M. Atrial fibrillation and mortality in African American patients with heart failure: results from the African American Heart Failure Trial (A-HeFT). Am Heart J. 2011 Jul;162(1):154-9. doi: 10.1016/j.ahj.2011.04.022. PMID 21742102